CLINICAL TRIAL: NCT06777472
Title: Clinical Study on Reducing Exacerbations of Asthma by Lung-benefiting Moxibustion Based on "Winter Disease Cured in Summer"
Brief Title: Clinical Study of Lung-benefiting Moxibustion Reduce Exacerbations of Asthma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cuiling Feng (Other)
Collaborators: The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Zhuhai Hospital of Integrated Traditional Chinese and Western Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Cuiling Feng, professor, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024PHB342-001
Record Dates: First submitted 2024-12-29; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Asthma
Keywords: asthma out of control; lung-benefiting moxibustion; Treating winter diseases in summer; RCT
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test group (Experimental): On the basis of the control group, lung-benefiting moxibustion treatment will be given.Details are as follows：
  1. The procedure of moxibustion includes 13 steps: selecting the body position, choosing the point, disinfecting, applying ginger juice, sprinkling moxibustion powder, covering mulberry paper, laying ginger mud, placing moxa cone, lighting moxa cone, changing moxa cone, removing ginger mud, gently rubbing moxibustion spot and placing blisters; The time of each application of moxibustion is 90 minutes.
  2. Treatment course: Start 10 days before the "early onset", once every 10 days, intervene 5 times, 1 year as one cycle, 2 consecutive cycles.
  Interventions: Other: lung-benefiting moxibustion; Drug: The specific drug comes from "GINA (2024)"
- control group (Active Comparator): Refer to "GINA (2024)". Regulations on combined medication: When complications occur during treatment, symptomatic treatment can be given according to the clinical situation. At the same time, the name, manufacturer, batch number, usage, dosage, course of treatment, etc. of the drug should be recorded in detail.
  Interventions: Drug: The specific drug comes from "GINA (2024)"

INTERVENTIONS:
Other: lung-benefiting moxibustion — A kind of external treatment，the treatment theory is to treat winter diseases in summer.
  Arms: test group
Drug: The specific drug comes from "GINA (2024)" — Refer to "GINA (2024)".

SUMMARY:
For patients with poor asthma control, on the basis of treatment guided by GINA guidelines, lung-benefiting moxibustion treatment will be given, and it will be applied 10 days before "early onset", once every 10 days, and the follow-up was 45 weeks, 1 cycle per year, for 2 consecutive cycles (2 years). The annual number of flare-up of asthma patients will be used as the main outcome index to evaluate the clinical effect of lung-benefiting moxibustion on reducing exacerbations of asthma. By observing immunoglobulin, T cell subsets and other indicators, the advantage population and mechanism of moxibustion in treating patients with poor asthma control will be clarified.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnosis of asthma (remission);
* Patients with poor clinical control;
* Age 18-80 years old;
* Voluntarily undergo treatment and sign an informed consent form;

Exclusion Criteria:

* Patients combined with pulmonary abscess, pulmonary fibrosis, active pulmonary tuberculosis, bronchiectasis or other lung diseases;
* Patients with severe cardiovascular and cerebrovascular diseases (malignant arrhythmia, unstable angina pectoris, acute myocardial infarction, cardiac functional classification≥III, stroke, cerebral hemorrhage, etc.)；
* Patients with severe liver diseases (liver cirrhosis, portal hypertension, bleeding due to esophageal and gastric varices, etc.) or severe kidney diseases (renal dialysis, kidney transplantation, etc.)；
* Patients with confusion, various mental disorders, etc., who are unable to communicate normally;
* Pregnant and lactating women;
* Patients with heat phlegm pattern through TCM pattern differentiation；
* Patients participating in other clinical trials within 1 month prior to enrollment;
* Received TCM external treatment such as lung-benefiting moxibustion for 1 year;
* Patients allergic to moxibustion drugs, smoke, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Annual number of flare-up of asthma | 1year
  Frequency

SECONDARY OUTCOMES:
ACT and ACQ questionnaires | Before treatment, and at 7, 13, 26, 39, 52, 59, 65, 78, 91, and 104 weeks.
  1. ACT asthma control test A score of 25 indicates well-controlled asthma, 20-24 indicates partially controlled asthma, and 20 indicates uncontrolled.
  2. Asthma Control Questionnaire <0.75 points indicates that asthma is completely controlled: 0.75-1.5 points indicates good control of asthma: >.15 points indicates that asthma is not well controlled
AQLQ scale | Before treatment, and at 7, 13, 26, 39, 52, 59, 65, 78, 91, 104 weeks.
  Asthma Quality of Life Questionnaire When calculating the overall score, the scores of each dimension are averaged to obtain a score between 0 and 7. The higher the score, worse the patient's quality of life. According to the AQLQ scoring criteria, a score above 5 indicates a relatively good quality of life, while a below 3 indicates a poor quality of life.
Pulmonary ventilation test and Diastolic test | Pulmonary ventilation test will be performed once before treatment,and at 52, 104 weeks.Diastolic tests will be performed once before treatment.
  Ventilation function test ml
FeNO | Before treatment,and at 52, 104 weeks.
  The fractional concentration of exhaled nitric oxide
Eosinophils count,Serum total IgE,and T-Lymphocyte Subsets | Before treatment,and at 7, 52, 59, 104 weeks.
  EO# x 10^9/L Ig E IU/mL percent of CD4+ cell、CD8+ cell 、CD4+/CD8+ cell

IPD SHARING:
Plan to Share IPD: Undecided
have not decided